CLINICAL TRIAL: NCT02340871
Title: Finding Genes With NGS Techniques in Whom Mutations Cause Neurological Diseases
Acronym: NGS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Charite University, Berlin, Germany (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0643-13; 1ZIAAG000958-12 (NIH)
Record Dates: First submitted 2015-01-06; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2014-12

CONDITIONS: Neurological Diseases
Keywords: Neurogenetics; genetic testing
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Genetic Neurological Diseases: The group consists of patients with a neurological disease that are tested for finding the genetic basis of their disease.The neurological signs and symptoms include ataxia, intellectual disability, seizures, movement disorders, migrational disorders, macrocephaly, microcephaly and various other signs and symptoms. The group consists of patients from 1-year-old until 90 years who are having a neurological disease as stated above or who are the parents or siblings of the affected patients. Blood specimens will be taken from them and DNA will be extracted for next generation studies like whole exome sequence or whole genome sequence. This process is called genetic testing. The current proposal will assist in diagnosing children and families with a neurological disease for genetic counseling.
  Interventions: Genetic: Genetic testing

INTERVENTIONS:
Genetic: Genetic testing — Patients suspected of harboring a genetic neurological disease will be summoned to take a blood test. DNA will be extracted from the blood and sent to the collaborating hospital labs for next generation sequencing.

SUMMARY:
In Israel, because of special qualification in neurogenetics, during a 30 year career ,we have found, characterized and treated at least 13 novel neurological diseases. The genetic basis was elucidated with geneticist colleagues both in Israel and worldwide. The diseases we have found encompass all the fields of pediatric neurology including intellectual disability, epilepsy, muscle-nerve disorders, malformations of the brain, microcephaly, macrocephaly, cerebellar ataxia, chorea. dystonia, cerebral palsy and many other symptoms and signs.

We are especially interested in consanguineous families, in whom the parents are first or second degree cousins. These families often bear autosomal - recessive diseases. If the family is informative - with 2 or more affected children - then with current genetic techniques there is a good chance of finding the causative gene to this specific disease. This is not only a theoretical - academic accomplishment. In practice, after discovering the gene, the family is given genetic counseling and in their further pregnancies the geneticists will examine either by preimplantation genetic diagnosis (PGD) or amniocentesis if the embryo is affected or not. In the early stages of the pregnancy if the embryo is indeed affected by the disease caused by the gene we have found and the religious official consents, genetic counseling can offer termination of pregnancy to the couple.

Needless to say, we know the immense burden of an affected child on the family, community and society. The parents are guilt-ridden, the affected child draws extensive resources from educational, health and rehabilitation authorities. We can contribute to the well-being of the family and the clan (because many times the relatives are affected).

We can perform sophisticated genetic studies such as Whole Genome Sequencing and Whole Exome Sequencing.After an informative family is recruited to the study, we will explain the aims of the research. The parents and eligible patients will sign informed consent forms, according to the local Helsinki Board. Blood samples will be taken in Israel, DNA extracted in the Israeli lab and then shipped coded to the researchers in USA or Germany. If the researchers will find a new gene the family will be notified and given appropriate genetic counseling. We will continue to follow and treat the family onwards.

DETAILED DESCRIPTION:
In Israel there are various sub-populations with a tendency to consanguinity. Among them are the Arab-Muslim, Druze, Bedouin, Sephardi Jews and to a lesser extent Ashkenazi Jews.

Consanguinity (especially between 2 first cousins) exposes the couple to various genetic diseases at a risk of 25% per each pregnancy. This phenomenon is based on Mendelian autosomal-recessive inheritance. When the couple is from the same family or clan, or even from the same ethnic origin , there is a probability that "dormant" abnormal genes will pass through generations of intermarriage, thus rendering the couple as "carriers" and producing a risk of 25% for the offspring to be affected.

Many of the autosomal-recessive diseases have neurological features such as : developmental delay, intellectual disability, epilepsy and motor and/or sensory impairment. These diseases carry a heavy burden on the family, community and the educational, health and welfare authorities. The disabled children are often handicapped, go to special education programs, are not independent in daily living tasks, are often sick and in need of hospitalization. They will grow up needing special housing facilities. Their life span is usually shorter than normal. These children are dependent on their parents, they subdue the parents to misery, interparental conflicts and susceptibility to divorces. Most of the neurological diseases are untreatable nowadays. Most of the medical effort focuses on their prevention. For example, by finding the gene for a specific neurological condition, we could search for that same gene in the couple's next pregnancy. If the fetus is found to be affected we could offer genetic counseling and a possibility of pregnancy termination and so the family avoids the birth of an affected sibling.

When an individual with a neurogenetic disease is enrolled to the study a careful history is taken to characterize the neurological syndrome, to see if other family members are affected by the same condition, and a pedigree is drawn. We compare the neurological signs and symptoms to information data webs like " PUBMED" or "Online Mendelian Inheritance in Man", and if we don't find a similar description we refer to the family as harboring a new disease with a novel gene.

We work with neurogenetic colleagues abroad like Dr. Andy Singleton in National Institute of Aging, NIH, U.S.A of Dr. Markus Schuelke from Charite Hospital, Berlin, Germany.

We take on ourselves to search for the families, explain to them what are the purposes of the research and their consequences. If we suspect a new gene, we will ask the parents or patients to sign informed consent forms according to our approved Helsinki board. We will take a sample of 10 cc blood in order to extract DNA. The DNA will be extracted in the genetic lab in Israel. A coded DNA will be sent to the researcher abroad. After 12 years the sample will be returned coded to the lab in Israel.

The researchers abroad will use homozygosity mapping techniques as well as NEXT GENERATION SEQUENCING like WHOLE EXOME SEQUENCING and WHOLE GENOME SEQUENCING.

If a new gene is found we will arrange for proper genetic counseling and explain the implications of the genetic data on the individual and his family. We will provide the family with symptomatic or palliative further therapy as needed.

ELIGIBILITY:
Inclusion Criteria:All patients with neurological conditions, their siblings and parents. -

Exclusion Criteria:None

-

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a constellation of neurological findings that seem to be a new syndrome or disease are enrolled to the study to decipher the genetic basis of their disease with next generation techniques.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
75 patients with a neurological disease will be tested by Next Generation Sequence techniques to find a genetic basis for their disease | 3 years
  The outcome (the finding of a new gene will be reported to the patient and his caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Straussberg, M.D, Principal Investigator — Schneider's Children Medical Center
Locations (1):
- Scneider's Children Medical Center, Petah Tikva, Israel